CLINICAL TRIAL: NCT05850793
Title: Comparison of Progressive Motor Imagery and Sensorimotor Exercises in Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Comparison of Progressive Motor Imagery and Sensorimotor Exercises in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ebru gulek karaduz, Physiotherapist (MSc ) / PhD (continous) / Lecturer Ebru Gülek Karadüz, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ebrugk
Record Dates: First submitted 2023-03-18; First posted 2023-05-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis, Knee
Keywords: rehabilitation; motor imagery training; sensorimotor training; balance; functional performance
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and the researcher who evaluated the analysis are blind to the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sensorimotor Exercise Training (Experimental): Sensorimotor exercise content has been prepared based on previous sensorimotor, balance and proprioceptive studies in the literature. It is organized as a structured traditional exercise program + SM training content.
  Interventions: Behavioral: Sensorimotor Exercise; Behavioral: Conventional Exercise
- Progressive Motor Imagery Training (Experimental): In order to sequentially activate the cortical motor networks and improve cortical organization, a literature-supported program including the components of AMI training (first stage laterality training, second stage motor imagery and third stage mirror therapy) was prepared and a six-week structured exercise program suitable for knee joint treatment + AMI training was prepared.
  Interventions: Behavioral: Conventional Exercise; Behavioral: Progressive Motor Imagery Exercise
- Conventional Exercise Training (Active Comparator): A 6-week program was prepared from traditional treatment exercises based on previous studies in knee osteoarthritis. It consists of progressive muscle strengthening of Quadriceps, Hamstrings and gluteals and also stretching exercises.
  Interventions: Behavioral: Sensorimotor Exercise; Behavioral: Conventional Exercise; Behavioral: Progressive Motor Imagery Exercise

INTERVENTIONS:
Behavioral: Sensorimotor Exercise — Balance, perturbation , aging and strengthing exercise will be performed for knee
  Arms: Conventional Exercise Training; Sensorimotor Exercise Training
Behavioral: Conventional Exercise — Range of motion, strengthing and stretching exercise will be performed for knee
  Other Names: traditional exercise for osteoarthritis
Behavioral: Progressive Motor Imagery Exercise — Different types of exercises will be applied targeting muscle strength, proprioceptive sense or brain neurons for knee
  Arms: Conventional Exercise Training; Progressive Motor Imagery Training

SUMMARY:
Osteoarthritis is the most common type of arthritis, which can affect all joints in the body and includes synovial inflammation, cartilage degeneration, osteophyte formation and bone remodeling in its pathophysiology. Many approaches are used in its treatment, and the effectiveness of exercise in conservative treatment has been proven. Many exercise methods such as strengthening, balance, aquatherapy are applied, but there is no definite consensus on exercise prescribing.Programs that focus on restoring balance and proprioception are called "sensorimotor or neuromuscular trainings". Previous studies have shown that neuromuscular exercises reduce pain, improve function, improve balance, and cause positive biomechanical changes in knee osteoarthritis and meniscus injuries. Progressive Motor Imagery (AMI) is an approach in rehabilitation where the focus is on progressive brain exercise. It is an education that approaches patients with pain, activity limitation and functional loss with a holistic view within the framework of the biopsychosocial model.

The aim of this study; to examine the effects of two current treatment programs (AMI, SM training) on symptoms, functionality, balance and proprioception parameters in osteoarthritis rehabilitation.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common arthritis, affecting more than 300 million adults worldwide. The pathophysiology of OA, which can affect all joints in the body, includes synovial inflammation, cartilage degeneration, osteophyte formation, and bone remodeling. These changes in OA, a chronic and degenerative joint disease, impair joint stability and function, causing pain. With the deterioration of the dynamic balance between production and destruction in the articular cartilage and subchondral bone, the joint becomes unable to meet the load . The knee joint is the most commonly affected joint in the body by OA; it also ranks eleventh among the leading causes of global disability. Typically, patients with knee OA experience pain, swelling, decreased muscle strength (especially the quadriceps femoris), joint stiffness, and loss of function

Therapeutic exercise, weight control in obese patients, self-efficacy and self-management programs, use of orthoses, topical and oral nonsteroidal anti-inflammatory drugs, intra-articular injections, radiofrequency and surgical methods are used in the management of knee OA. The primary treatment in the treatment of OA is to prefer conservative practices such as exercise and education .

Progressive Motor Imagery (AMI) is an approach in rehabilitation where the focus is on progressive brain exercise. It is an education that approaches patients with pain, activity limitation and functional loss with a holistic view within the framework of the biopsychosocial model. It consists of three components in turn: Laterality training (left-right discrimination training), motor imagery (imagining movements), and the third step mirror therapy (providing visual feedback through the mirror). Laterality (closed imagery) is the process of determining whether a limb is a left or right limb, or that the patient is turning right or left for the spine. Motor imagery (open imagery) is the patient's internal, external and kinesthetic imagining of their movements and postures. Mirror therapy (visual feedback) refers to the use of a mirror to present an inverted image of a limb, thereby tricking the brain. By following these three steps, it is aimed to sequentially activate cortical motor networks and improve cortical organization.

* The aim of our study; to examine the effects of two current treatment programs (AMI, SM training) on symptoms, functionality, balance and proprioception parameters in osteoarthritis rehabilitation.
* The study is a prospective, three arm ,randomized controlled trial. A total participant number was calculated with Gpower as 54 patients with %90 power.
* There will be 3 groups and participants will perform the exercises which included their group 2 times a week for 6 weeks, accompanied by a physiotherapist.Each group includes 18 patients.
* Evaluations will be made at the start of treatment, at 6th weeks and 12th weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee OA according to the criteria of the American Society of Rheumatology (ACR),
* Stage 2 or 3 according to Kellgren Lawrence radiological staging criteria,
* Between the ages of 50 and 65,
* Body mass index below 35 kg/m²,
* Pain intensity defined by the patient in the last 3 months is at least 3 out of 10 according to NPRS,
* There are no obstacles to being included in the exercise program,
* Patients with a score of at least 24 on the Standardized Mini Mental Test will be included.

Exclusion Criteria:

* Receiving any physiotherapy program or injection treatment in the last 3 months,
* Having a diagnosis of additional pathology other than OA in the knee, having a history of knee injury / surgery in the past
* Having uncontrollable hypertension, cardiovascular and neurological diseases that will prevent exercise,
* The patient has any vision, hearing or cognitive problems that will prevent him from complying with the treatment,
* Providing ambulation with an assistive device

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Balance | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th weeks
  For balance and fall risk assessment, the Biodex Balance System (BBS) (Biodex Medical Systems, Inc. 20 Ramsey Road, Shirley, New York) will be used. Computer result will be used to see falling risk and stability postural problems as anteroposterior and mediolateral.
  In the evaluation, while the patient stands without shoes on the BBS platform, the patients are asked to place their feet on the marked place, hold the BBS monitor and focus. The patient is asked to keep the cursor on the screen in the smallest circle shown on the device screen for 20 seconds while applying surface movements that can move between 20 and 360 degrees that will disrupt postural stability at different levels (12 most stable, 1 most mobile). Based on previous studies, the static assessment will be assessed at level 12, and the dynamic assessment and risk of falling will be assessed at level 8.

SECONDARY OUTCOMES:
Pain of joint | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th week
  The Numerical Rating Pain Scale (NPRS) is frequently used to measure and monitor the severity of pain. Absence of pain is defined by 0 and excruciating pain by 10.
Proprioception | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th week
  The passive-active angle repetition test is often preferred to evaluate proprioception. In this test, the knee is moved (actively or passively) toward a specified target angle with the patient's eyes open. After a few seconds, the knee is returned to the starting position and the target angle is repeated. Following this, the patient is asked to reconstruct the perceived angle with the same knee while his eyes are closed, and how much the knee joint deviates from the target angle is calculated. The error will be recorded as deviated angle .

OTHER OUTCOMES:
Functional Evaluation | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th week
  The Western Ontario and McMaster Universities Osteoarthritis Index; It was developed specifically for OA in order to determine the physical function levels of patients based on their own reports. In the literature, it is seen that the WOMAC score is frequently used to evaluate the functional status of daily life in patients with OA. Translation of WOMAC into Turkish, validity and reliability studies were carried out. In the scale consisting of 24 questions and 3 subsections, the first section evaluates pain (5 questions), the second section evaluates joint stiffness (2 questions), and the third section evaluates the level of difficulty experienced by the patient while performing physical functions (17 questions). The scale scores is reported between 0 to 100 point and high scores show worse outcome..
Range of Motion | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th week
  Goniometric measurement is an objective method that is frequently used in the evaluation of joint range of motion (ROM). Universal goniometer will be used for all measurements in the study. Flexion and extension ROM measurements of both knee joints will be measured in all patients, and arithmetic mean values will be recorded by repeating each measurement three times. The result will be record as angle.
Cognitive status | only at baseline evaluation for inclusion criteria (MMSE ≥ 24 point)
  Cognitive status assessment will be made using the Standardized Mini Mental Test (Mini Mental State Examination, MMSE). It is a test consisting of 30 questions and evaluated over 30 points, providing data about cognitive status by evaluating cognitive functions such as orientation, memory, calculation, speaking, and drawing a complex polygon. High Scores shows better cognitive status.
Mobility | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th week
  The Timed Up and Go Test is a test used to evaluate the mobility of the patient. It measures the time it takes for a participant to stand up from a comfortable 45-cm-high chair, walk 3 meters quickly, cross the line on the floor, turn, walk back to the chair, and sit down. The participant is encouraged to do the test very quickly. High scores shows worse outcome.
Lateralization | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th week
  Lateralization will be evaluated with the Recognise™ application developed by the "Neuro Orthapaedic Institute". Recognise™ is a valid and reliable application used to measure lateralization speed and accuracy (37). Separate applications have been developed for neck, waist, knee, foot, shoulder and hand. Application result will be used as accuracy rates (%) and speed as time.
Patient Satisfaction | change from baseline to posttreatment 6th weeks , change from posttratment 6th weeks to 12th week
  Patient satisfaction will be evaluated with the Global Rating of Change (GRC) as a score between -2 to 2 point. Lower score shows worse satisfaction outcome.

CONTACTS AND LOCATIONS:
Overall Officials: EBRU KARADÜZ, PhD(c), Principal Investigator — İstanbul Medipol University; Sena TOLU, Asist Prof, Study Chair — Medipol Mega Hospital; Candan Algun, Prof, Study Chair — İstanbul Medipol University
Locations (1):
- Ebru Karadüz, Fatih, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Busija L, Bridgett L, Williams SR, Osborne RH, Buchbinder R, March L, Fransen M. Osteoarthritis. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):757-68. doi: 10.1016/j.berh.2010.11.001. PMID 21665124
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Sharma L. Osteoarthritis of the Knee. N Engl J Med. 2021 Jan 7;384(1):51-59. doi: 10.1056/NEJMcp1903768. No abstract available. PMID 33406330
- [Background] Zhang W, Doherty M, Peat G, Bierma-Zeinstra MA, Arden NK, Bresnihan B, Herrero-Beaumont G, Kirschner S, Leeb BF, Lohmander LS, Mazieres B, Pavelka K, Punzi L, So AK, Tuncer T, Watt I, Bijlsma JW. EULAR evidence-based recommendations for the diagnosis of knee osteoarthritis. Ann Rheum Dis. 2010 Mar;69(3):483-9. doi: 10.1136/ard.2009.113100. Epub 2009 Sep 17. PMID 19762361
- [Background] Dominguez-Navarro F, Igual-Camacho C, Silvestre-Munoz A, Roig-Casasus S, Blasco JM. Effects of balance and proprioceptive training on total hip and knee replacement rehabilitation: A systematic review and meta-analysis. Gait Posture. 2018 May;62:68-74. doi: 10.1016/j.gaitpost.2018.03.003. Epub 2018 Mar 5. PMID 29525292
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controlled trial. Neurology. 2006 Dec 26;67(12):2129-34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID 17082465
- [Background] Baird CL, Sands L. A pilot study of the effectiveness of guided imagery with progressive muscle relaxation to reduce chronic pain and mobility difficulties of osteoarthritis. Pain Manag Nurs. 2004 Sep;5(3):97-104. doi: 10.1016/j.pmn.2004.01.003. PMID 15359221
- [Result] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149